CLINICAL TRIAL: NCT05924997
Title: A Phase Ib/II Trial Evaluating the Efficacy and Safety of Adebrelimab, Camrelizumab Plus Apatinib as First-line Therapy in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Adebrelimab, Camrelizumab Plus Apatinib as First-line Therapy in Patients With Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-514-01
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: adebrelimab; camrelizumab; apatinib; hepatocellular carcinoma; first-line therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental)
  Interventions: Drug: adebrelimab, camrelizumab plus apatinib

INTERVENTIONS:
Drug: adebrelimab, camrelizumab plus apatinib — adebrelimab (RP2D, Q3W)+ camrelizumab 200mg Q3W+ apatinib 250mg qd, with 3 weeks (21 days) as a treatment cycle

SUMMARY:
This is a prospective, single-arm, phase Ib/II trial . The objective of this study is to evaluate the efficacy and safety of adebrelimab, camrelizumab plus apatinib as first-line therapy in patients with advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
This study is divided into two stages: in the Ib stage, the tolerance and safety of adebrelimab, camrelizumab plus apatinib in the treatment of patients with advanced solid tumors were studied; The second phase is a single-arm, open and multi-center clinical study. The improvement of objective response rate (ORR) in patients with advanced HCC by first-line treatment with adebrelimab, camrelizumab plus apatinib was observed and evaluated.

■ The first stage

In order to effectively investigate the safety of adebrelimab, camrelizumab plus apatinib in the treatment of patients with advanced solid tumors, the following cohort (dose level) studies are planned:

Queue 1: adebrelimab 10mg/kgQ3W+ camrelizumab 200mgQ3W+ apatinib 250mgqd. Queue 2: adebrelimab 20mg/kgQ3W+ camrelizumab 200mgQ3W+ apatinib 250mgqd. Using i3+3 design, 3~6 subjects are expected to be enrolled in each cohort. Every 3 weeks (21 days) is a treatment cycle, and DLT observation period is the first and second cycles of combined administration. After passing the safety evaluation of DLT observation period, the next dose group experiment can be gradually entered.

■ The second stage According to the results of the first phase, the recommended dose of phase II study (RP2D) was selected for further efficacy and safety evaluation in patients with advanced hepatocellular carcinoma who had not received systematic treatment before.

The objective remission rate (ORR) was the main end point of the study, and 46 subjects were planned to be enrolled. After fully knowing and signing the informed consent form, the subjects will receive the study treatment: adebrelimab (RP2D, Q3W)+ camrelizumab 200mgQ3W+ apatinib 250mgqd, with 3 weeks (21 days) as a treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered to join this study and signed informed consent;
* ≥ 18 years old (calculated on the day of signing the informed consent), both men and women can be used;
* Patients with advanced or metastatic solid tumor confirmed by histology or cytology (stage Ⅰb); Patients with hepatocellular carcinoma diagnosed by EASL/AASLD diagnostic criteria, histopathology or cytology are not suitable for surgery or local treatment, or progress after surgery and/or local treatment (stage II);
* Subjects must be able to provide fresh or archived tumor tissues (formalin-fixed, paraffin-embedded [FFPE] tissue blocks or at least 5 unstained FFPE slides) and their pathological reports. If the subjects can provide less than 5 unstained slides or the tumor tissue is unavailable (for example, because of previous diagnostic tests), after discussion, they may be allowed to join the group according to the specific circumstances;
* For patients who have progressed after local treatment, local treatment (including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) has been completed at least 4 weeks before the baseline imaging scan, and the toxic reactions caused by local treatment (except alopecia) must be restored to the fifth edition of the National Cancer Institute-General Terminology Standard for Adverse Events (NCI-CTCAEV 5. 0) rating ≤1 level;
* Never received any systematic treatment for HCC before;
* There is at least one measurable lesion (according to the requirements of RECISTv1.1, the long diameter of the measurable lesion in spiral CT scanning is ≥10mm or the short diameter of swollen lymph nodes is ≥ 15 mm; Lesions that have received local treatment in the past can be used as target lesions after definite progress according to RECISTv1.1 standard);
* Child-Pugh liver function classification: A or B)
* The score of physical condition of the Eastern Cancer Cooperative Group (ECOG) is 0 ~ 2;
* The expected survival time is ≥12 weeks;
* The functions of major organs are basically normal, with serious dysfunction of blood, heart, lung, liver, kidney, bone marrow and immunodeficiency diseases, which meet the requirements of the scheme: a) Routine blood examination: (Except hemoglobin, no blood transfusion within 14 days before screening, no use of granulocyte colony-stimulating factor [G-CSF] and no use of corrective treatment within 7 days) i. Hemoglobin ≥ 90g/L. Ii. Neutrophil count ≥ 1.5× 109/L; Iii. Platelet count ≥ 50× 109/L; B) Biochemical examination: (albumin was not transfused within 14 days) i. Serum albumin ≥ 29g/L; Ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 times the upper limit of normal value (ULN); Iii. Total bilirubin (TBIL)≤1.5 times ULN；; Iv. Creatinine Cr≤1.5 times ULN or Cr clearance rate > 50mL/min(Cockcroft-Gault formula is as follows) Male: Cr clearance rate =((140- age) × body weight) /(72× blood Cr) Female: Cr clearance rate =((140- age) × body weight)/(72 Blood Cr unit: mg/ml; V. Urine protein < 2+ (if urine protein ≥2+, 24-hour (h) urine protein quantification can be performed, and 24-hour urine protein quantification < 1.0g can be enrolled); C) Coagulation function: APTT and INR)≤1.5×ULN (for anticoagulant therapy with stable dosage such as low molecular weight heparin or warfarin and INR can be screened within the expected therapeutic range of anticoagulant); D) thyroid stimulating hormone (TSH) ≤ ULN; If abnormal, T3 and T4 levels should be investigated, and normal T3 and T4 levels can be selected; E) Color Doppler echocardiography: Left ventricular ejection fraction (LVEF) is greater than or equal to 60%.
* If the patient suffers from active hepatitis B virus (HBV) infection: the HBV- deoxyribonucleic acid (DNA) must be less than 2× 103 IU/ml and he is willing to receive antiviral treatment (according to local standard treatment, such as entecavir) during the study period, and the doctor will judge whether the patient is eligible for enrollment according to the individual situation of the patient under the condition of monitoring the virus copy number; Hepatitis C virus (HCV) ribonucleic acid (RNA) positive patients must receive antiviral treatment according to local standard treatment guidelines, and their liver function should be within the level 1 increase of CTCAE1.
* Fertile women: they must agree to abstain from sex (avoid heterosexual intercourse) or use reliable and effective methods of contraception for at least 120 days from the signing of the informed consent form to the last administration of the study drug. And the serum HCG test must be negative within 7 days before the start of the study treatment; And must be non-lactating. If a female patient has menstruated, has not yet reached the post-menopausal state (continuous non-menstrual period ≥12 months, and no other reasons have been found except menopause), and has not received sterilization surgery (such as hysterectomy, bilateral tubal ligation or bilateral oophorectomy), it is considered that the patient has fertility.
* For male patients whose partner is a woman of childbearing age, they must agree to abstain from sex for at least 120 days from signing the informed consent form until the last administration of the study drug, or to use reliable and effective methods for contraception. Male subjects must also agree not to donate sperm during the same period. Male subjects whose partners are pregnant must use condoms, and no other contraceptive methods are needed.

Exclusion Criteria:

* Cholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and fibreboard cell carcinoma; Have other active malignant tumors except HCC within 5 years or at the same time. Localized tumors that have been cured, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ, breast cancer in situ, etc., can be included in the group;
* Patients who are ready to undergo or have previously received an organ or allogeneic bone marrow transplantation;
* Received other experimental drugs within 28 days before starting the study treatment;
* Moderate and severe ascites with clinical symptoms requires therapeutic puncture, drainage or Child-Pugh score > 2 (except for those who only show a small amount of ascites on imaging but are not accompanied by clinical symptoms); Uncontrolled or moderate or above pleural effusion and pericardial effusion;
* Patients who have a history of gastrointestinal bleeding or have a clear tendency of gastrointestinal bleeding within 6 months before the start of the study and treatment, such as: bleeding-risk or severe esophageal and gastric varices, local active gastrointestinal ulcer lesions, and persistent fecal occult blood positive, can not be included in the group (if the fecal occult blood is positive in the baseline period, it can be rechecked, if it is still positive after the recheck, it needs to undergo gastroduodenoscopy (EGD), and if the EGD indicates bleeding-risk esophageal and gastric varices, it can not be included).
* Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the start of the study treatment;
* Known hereditary or acquired bleeding (such as coagulation dysfunction) or thrombotic tendency, such as hemophilia patients; At present, or in the near future (within 10 days before the start of the study treatment), full-dose oral or injection anticoagulants or thrombolytic drugs have been used for therapeutic purposes (low-dose aspirin and low-molecular-weight heparin are allowed for preventive use);
* Aspirin (> 325mg/ day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel and cilostazol are currently being used or recently used (within 10 days before the start of the study treatment);
* Thrombosis or embolism occurred within 6 months before the start of the study, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction) and pulmonary embolism;
* There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) Cardiac insufficiency above Grade II according to the standards of new york Heart Association (NYHA) or cardiac color Doppler examination: LVEF (Left Ventricular Ejection Fraction) < 50%; (2) Unstable angina pectoris; (3) myocardial infarction occurred within one year before the start of study and treatment; (4) Clinically significant supraventricular or ventricular arrhythmia needs treatment or intervention; (5) QTc > 450 ms (male); QTc>470ms (female) (QTc interval is calculated by Fridericia formula; If the QTc is abnormal, it can be continuously detected for three times every 2 minutes, and the average value can be taken);
* Suffering from hypertension, which cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) (based on the average of BP readings obtained by ≥2 measurements), it is allowed to realize the above parameters by using antihypertensive therapy; Hypertensive crisis or hypertensive encephalopathy has occurred in the past;
* Major vascular diseases (for example, aortic aneurysm requiring surgical repair or recent peripheral artery thrombosis) occurred within 6 months before the start of study treatment; Severe, unhealed or split wounds and active ulcers or untreated fractures; Received major surgical treatment (except diagnosis) within 4 weeks before the start of the study treatment or expected major surgical treatment during the study period;
* Can't swallow pills, malabsorption syndrome or any condition that affects gastrointestinal absorption; Have suffered from intestinal obstruction and/or had clinical signs or symptoms of gastrointestinal obstruction within 6 months before the start of the study, including incomplete obstruction related to the original disease or requiring routine parenteral hydration, parenteral nutrition or tube feeding: At the initial diagnosis, patients with signs/symptoms of incomplete obstruction/obstruction syndrome/intestinal obstruction may be admitted to the study if they receive definite (surgical) treatment to relieve symptoms;
* There is evidence that there is pneumoperitoneum that cannot be explained by puncture or recent surgical operation;
* Past or present central nervous system metastasis; Metastatic diseases involving major airways or blood vessels (for example, portal vein trunk or vena cava that is completely occluded due to tumor invasion needs to be excluded from the group, portal vein trunk refers to the confluence of the splenic vein and superior mesenteric vein and the branch where hepatic portal vein divides into left and right branches) or large mediastinal tumor mass in the center (less than 30 mm from carina);
* Those with a history of hepatic encephalopathy; At present, patients with interstitial pneumonia or interstitial lung disease, or patients with a previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other subjects with pulmonary fibrosis, organized pneumonia (for example, bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or subjects with evidence of active pneumonia or severe impairment of lung function on chest computed tomography (CT) during the screening period are allowed to have radiation pneumonia in the radiation field. Active tuberculosis;
* Active autoimmune disease or history of autoimmune disease and possible recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects who can only be controlled by hormone replacement therapy can be included]); Subjects suffering from skin diseases without systematic treatment, such as vitiligo, psoriasis, alopecia, controlled type I diabetes treated with insulin or asthma in childhood have been completely relieved, and adults can be included without any intervention; Asthmatic patients who need bronchodilators for medical intervention cannot be included;
* Use immunosuppressant or systemic hormone therapy within 14 days before starting the study treatment to achieve the purpose of immunosuppression (the dose is > 10mg/ day of prednisone or other therapeutic hormones);
* Strong CYP3A4/CYP2C19 inducers used within 14 days before the start of study treatment include rifampicin (and its analogues) and Hypericum perforatum or strong CYP3A4/CYP2C19 inhibitors;
* It is known that there is a history of a severe allergy to any monoclonal antibody and anti-angiogenesis targeted drugs;
* Severe infection within 4 weeks before the start of study and treatment, including but not limited to hospitalization due to infection, bacteremia, or complications of severe pneumonia; Therapeutic antibiotics were given orally or intravenously within 2 weeks before the start of the study treatment (patients receiving preventive antibiotics (for example, patients who prevent urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible to participate in the study);
* patients with congenital or acquired immunodeficiency (such as HIV-infected people);
* Co-infection with hepatitis B and hepatitis C;
* Previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or previously received apatinib therapy;
* Patients have received live attenuated vaccine treatment within 28 days before the start of the study treatment, or expected to need such vaccine within 60 days after the last administration of adebelizumab.
* According to the researcher's judgment, the patient has other factors that may affect the study results or cause the study to be forced to terminate halfway, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory examination abnormalities, and family or society.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 2 years
  The proportion of subjects who achieved complete response (CR; all target lesions disappeared) or partial response (PR; the sum of the longest diameter of target lesions decreased by ≥ 30%) according to the RECIST1.1 standard.
Objective Response Rate | Up to approximately 2 years
  The proportion of subjects who achieved complete response (CR; the disappearance of any intratumoural arterial enhancement in all target lesions) or partial response (PR; at least a 30% decrease in the sum of the longest viable tumour diameters of target lesions) according to the mRECIST standard.
Adverse events (AEs) and serious adverse events (SAEs) | Up to approximately 2 years
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of adebrelimab, camrelizumab plus apatinib as first-line therapy in patients with advanced hepatocellular carcinoma.

SECONDARY OUTCOMES:
Progression Free Survival | Up to approximately 2 years
  The period of time from the start of treatment to progressive disease[PD] or death.
Duration of Response | Up to approximately 2 years
  The period of time from the days which achieved complete response [CR] or partial response[PR] to progressive disease[PD].
Disease Control Rate | Up to approximately 2 years
  The proportion of the sum of complete response [CR]、partial response [PR]、stable disease[SD] among the total cases.
Time to Progression | Up to approximately 2 years
  The period of time from the start of treatment to progressive disease [PD].
Overall Survival | Up to approximately 2 years
  The period of time from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No